CLINICAL TRIAL: NCT03308786
Title: HIV Reservoir Reduction With Interleukin-2
Acronym: IL2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: There were 3 instances of adverse events which were discussed with external safety monitoring committee and it was recommended that the study be terminated.
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Michael M. Lederman MD, Principal Investigator, Case Western Reserve University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AIDS 400: IL2
Record Dates: First submitted 2017-09-29; First posted 2017-10-13 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IL2 treatment (Experimental): Subcutaneous recombinant interleukin-2 (rIL2), 5 MIU twice daily for four consecutive days(cycle) every 8 weeks for 8 cycles, in addition to combination antiretroviral therapy.
  Interventions: Drug: Recombinant Interleukin-2

INTERVENTIONS:
Drug: Recombinant Interleukin-2 — Subcutaneous recombinant interleukin-2 (rIL2), 5 MIU twice daily for four consecutive days(cycle) every 8 weeks for 8 cycles
  Other Names: IL2, IL-2, rIL2, aldesleukin

SUMMARY:
The purpose of this pilot study is to examine the effects of eight 4-day cycles of subcutaneous recombinant interleukin-2 (rIL-2) given every 8 weeks on levels of replication-competent HIV in CD4 cells and on the size of HIV viral reservoir in up to 20 participants with chronically suppressed HIV infection (viral load <50 copies/mL).

DETAILED DESCRIPTION:
Interleukin-2 (IL-2) has been extensively studied in HIV infected individuals with no demonstrated clinical benefit as far as improving survival or decreasing risk of progression to AIDS. The results of the two landmark, international, multicenter, phase III, randomized trials of IL-2 in HIV infected participants (SILCAAT and ESPRIT) have been recently published. These trials, which started more than a decade ago, enrolled over 5800 participants who were randomized to anti-retroviral therapy (ART) +/- IL-2 and showed no benefit to IL-2 treatment in survival or progression to AIDS. Many individuals with HIV infection can lead normal lives on ART but replication-competent virus remains within resting CD4+ cells, referred to as the "HIV reservoir". There is a renewed interest in strategies to decrease or eliminate the viral reservoir in an attempt to provide a sterilizing or a functional "cure" for HIV that would allow the discontinuation of ART, which currently must be taken life-long. These therapies have long-term metabolic and cardiovascular toxicities as well as substantial cost. More recent data suggest that IL-2 administration may decrease the size of the HIV reservoir, getting ART-treated participants closer to levels of HIV persistence that may ultimately allow for sterilizing or functional cure.

The purpose of this pilot study is to examine the effects of eight 4-day cycles of subcutaneous recombinant interleukin-2 (rIL-2) given every 8 weeks on levels of replication-competent HIV in CD4 cells and on the size of HIV viral reservoir in up to 20 participants with chronically suppressed HIV infection (viral load <50 copies/mL).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed and dated by study participant.
2. Male or female, at least 18 years of age and not older than 65 years of age.
3. HIV-1 infection, documented by and FDA-approved ELISA, EIA, or rapid antibody detection method, and confirmed by a second approved antibody-based test or by a positive approved HIV RNA detection assay.
4. CD4+ T cell count ≥ 350 cells/mm3;
5. HIV-1 RNA < 50 copies/mL obtained within 60 days prior to study entry performed with an FDA-approved HIV-1 RNA assay.
6. Adequate venous access and no other contraindications for leukapheresis
7. Absolute neutrophil count (ANC) > 2000/mm3
8. Hemoglobin level >10 g/dL (males); > 9.5 g/dL (females)
9. Platelet count >150,000/mm3
10. Serum creatinine <1.5 mg/dL
11. AST and ALT <2.5 times the upper limit of normal
12. TSH, T3, and T4 levels within the normal range of the processing laboratory.
13. Anti-thyrosine peroxidase (TPO) within the normal range of the processing laboratory.
14. Willing to comply with study-mandated evaluations; including not changing antiretroviral regimen (unless medically indicated) during the study period.
15. All participants must have received HAART, and had viral loads below the limit of quantification of the assay for at least 1 year. Participants who had intermittent isolated episodes of detectable low-level viremia < 500 copies RNA/mL flanked by viral loads below the limit of quantification of the assay will remain eligible.
16. On a stable 3-drug combination antiretroviral regimen (no changes to treatment within 4 weeks of enrollment) and willing to continue on current antiretroviral therapy for the duration of the study, unless otherwise medically indicated. The study principal investigator can approve a 2-drug antiretroviral regimen on a case-by-case basis.

Exclusion Criteria:

1. Childbearing potential for female participants. For the purposes of this study, a woman is considered to be of childbearing potential if she is postmenarche, has not had a documented surgical sterilization procedure, has an intact uterus and at least 1 ovary, and has had a spontaneous menstrual period in the last 2 years.
2. Acute or chronic hepatitis C infection, defined as a positive plasma HCV RNA using any FDA-approved qualitative or quantitative test in a participant with a positive HCV antibody (HCV RNA testing is not required in participants with a negative HCV antibody). Participants who have completed a course of a direct-acting antiviral agent for hepatitis C and have a confirmed plasma HCV RNA level below the limit of detection of the assay 12 weeks or longer after completion of therapy will be eligible.
3. Acute or chronic hepatitis B infection, defined as a positive HBV surface antigen or a positive HBV DNA.
4. History of advanced chronic liver disease, including cirrhosis, advanced liver fibrosis, severe portal hypertension, or manifestations or hepatic failure.
5. History of malignant disease that is not considered to be surgically or medically eradicated or that has required any form of therapy in the past 5 years.
6. Current diagnosis of congestive heart failure of any severity, uncontrolled angina or uncontrolled arrhythmias.
7. History of chronic lung disease that has required pharmacologic treatment, oxygen supplementation, medical monitoring, or hospitalization in the previous year, or that is expected to cause persistent or recurrent pulmonary symptoms or impairment. Examples of the latter include but are not limited to chronic bronchitis, emphysema, and pulmonary fibrosis.
8. History or any features on physical examination indicative of a bleeding diathesis.
9. History or current diagnosis of thromboembolic disease, including deep vein thrombosis and pulmonary embolism, or family history of the same.
10. History of hypersensitivity to radiological contrast media or anticipated need for exposure to radiological contrast media during the study period.
11. Use of chronic corticosteroids, hydroxyurea, or immune-modulating agents (e.g., interleukin-2, interferon-alpha or gamma, granulocyte colony stimulating factors, etc.) within 30 days prior to enrollment.

    NOTE: Use of inhaled or topical steroids is not exclusionary.
12. Breast-feeding.
13. Use of aspirin, warfarin or any other antithrombotic or antiplatelet agent during the 2-week period prior to leukapheresis.
14. History of autoimmune disorders, including but not limited to Crohn's disease, scleroderma, thyroiditis, inflammatory arthritis, myasthenia gravis, glomerulonephritis, systemic lupus erythematous, and vasculitis.
15. Type 1 diabetes mellitus.
16. History of thyroid disease that has required antithyroid or thyroid hormone replacement therapy at any time in the past.
17. Current continued use, or anticipated continued medical indication for nephrotoxic agents, including but not limited to aminoglycosides and other potentially nephrotoxic antimicrobials, indomethacin, high scheduled doses of other NSAIDs, and lithium salts.

    NOTE: Low doses or limited duration of these agents (i.e., ≤14 days) is not exclusionary.
18. Current continued use, or anticipated continued medical indication for hepatotoxic agents, including but not limited to amiodarone, methotrexate, and anticonvulsants and antimicrobials with elevated hepatotoxic potential.

    NOTE: Low doses or limited duration of these agents (i.e., ≤14 days) is not exclusionary.
19. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
20. Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to study entry that in the judgement of the investigator may compromise study participation or pose additional risks to the participant.
21. Any other condition that, in the opinion of the clinical investigator or sponsor, might compromise any aspect of this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benigno Rodriguez, MD, Study Chair — Case Western Reserve University; Michael Lederman, MD, Study Chair — Case Western Reserve University
Locations (1):
- AIDS Clinical Trials Unit, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IL2 Treatment
Started | 9
Completed | 0
Not Completed | 9
Not completed — study terminated after discussion with Safety Monitoring Committee | 9

BASELINE CHARACTERISTICS:
Arm/Group | IL2 Treatment
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 49 [35 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
CD4+ T cell count ≥ 350 cells/mm^3 [Median (Full Range); unit: cells/mm^3] — Flow Cytometric measurement of circulating CD4 positive t-cells (CD4 t-cells)
  cells/mm^3 | 808 [478 to 1230]
HIV-1 RNA < 50 copies/mL obtained within 60 days prior to study entry [Count of Participants; unit: Participants] | 9
on stable 3-antiretroviral medications with no changes for at least 4 weeks [Count of Participants; unit: Participants] | 9

OUTCOME MEASURES:

1. Primary Outcome: Latent HIV Reservoir Change by QVOA
Description: Change in the number of infectious units per million resting CD4+ T cells (IUPM) from baseline to the end of study treatment, as measured by the Quantitative Viral Outgrowth Assay (QVOA).
Time Frame: 15 months
Population: No data was collected.
Arm/Group | IL2 Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Correlation of Latent Reservoir Measure by QVOA to Latent Reservoir Measure by Intact Proviral DNA.
Description: Correlation coefficient between measures of the latent HIV reservoir by QVOA and measures of the latent HIV reservoir by the intact proviral DNA assay.
Time Frame: 15 months
Population: No data was collected.
Arm/Group | IL2 Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Correlation of Latent Reservoir Measure by QVOA to Latent Reservoir Measure by the Tat-rev Inducible Limiting Dilution Assay (TILDA).
Description: Correlation coefficient between measures of the latent HIV reservoir by QVOA and measures of the latent HIV reservoir by the Tat-rev inducible limiting dilution assay (TILDA).
Time Frame: 15 months
Population: No data was collected.
Arm/Group | IL2 Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Correlation of Latent Reservoir Measure by QVOA to Latent Reservoir Measure by the Envelope Detection by Induced Transcription-based Sequencing (EDITS)
Description: Correlation coefficient between measures of the latent HIV reservoir by QVOA and measures of the latent HIV reservoir by the Envelope Detection by Induced Transcription-based Sequencing (EDITS).
Time Frame: 15 months
Population: No data was collected.
Arm/Group | IL2 Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: In Vivo Induction of HIV Expression in Vivo as Measured by the Envelope Detection by Induced Transcription-based Sequencing (EDITS)
Description: Number of inducible cell-associated HIV mRNA copies per million CD4+ T cells at the beginning and end of rIL2 cycles 1, 4, and 8.
Time Frame: 15 months
Population: No data was collected.
Arm/Group | IL2 Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Plasma HIV RNA During rIL2 Exposure
Description: Plasma HIV RNA copies/mL by PCR at the beginning and end of rIL2 cycle 1.
Time Frame: baseline, day 7
Measure: Mean (Standard Deviation); unit: RNA copies/mL
Arm/Group | IL2 Treatment
Number analyzed (Participants) | 9
RNA copies/mL
  baseline | 10 (0)
  day 7 | 298 (522)

7. Secondary Outcome: Natural Killer (NK) Cell Phenotype During rIL2 Exposure
Description: Change in the percent of NK cells expressing CD16+CD56+ by flow cytometry from baseline to the end of study treatment.
Time Frame: baseline, day 7
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | IL2 Treatment
Number analyzed (Participants) | 9
percentage of cells
  baseline | 28.8 [19.8 to 37.5]
  day 7 | 35.8 [30.9 to 39.2]

8. Secondary Outcome: Natural Killer (NK) Cell Phenotype During rIL2 Exposure
Description: Change in the percent of NK cells expressing CD56+CD16- by flow cytometry from baseline to the end of study treatment.
Time Frame: baseline, day 7
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | IL2 Treatment
Number analyzed (Participants) | 9
percentage of cells
  baseline | 4.5 [3.1 to 5.2]
  day 7 | 12.7 [8.3 to 17.1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected until the study was terminated. This period was the time between enrollment into the study and study termination. The duration ranged from 8.3 months to 14.6 months,.
Description: Total number of participants at risk for All-Cause Mortality is 9. All-Cause mortality was zero.
Arm/Group | IL2 Treatment
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 2/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IL2 Treatment (N=9)
suspected capillary leak syndrome (Vascular disorders) | 1 (1) — grade 3 rash with hypotension and edema
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IL2 Treatment (N=9)
biochemical hypothyroidism (Endocrine disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
On the basis of recommendation of the SMC, the study was terminated. Because of this, the primary objective could not be achieved and most of the secondary objectives could not be achieved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT03308786/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT03308786/ICF_001.pdf